CLINICAL TRIAL: NCT07319481
Title: Preliminary Effectiveness and Feasibility of Transcutaneous Acupoints Electrical Stimulation on Chemotherapy-induced Peripheral Neuropathy Among Chinese Children With Acute Lymphoblastic Leukemia: A Randomized Controlled Trial
Brief Title: Preliminary Effectiveness and Feasibility of Transcutaneous Acupoints Electrical Stimulation on Chemotherapy-induced Peripheral Neuropathy Among Children With Acute Lymphoblastic Leukemia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: The Affiliated Cancer Hospital of Zhengzhou University & Henan Cancer Hospital (Unknown)
Responsible Party: Principal Investigator, Dr Eva Ho, Associate professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Electrical stimulation
Record Dates: First submitted 2025-12-21; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Chemotherapy Induced Peripheral Neuropathy (CIPN)
Keywords: acute lymphoblastic leukemia; transcutaneous acupoints electrical stimulation; children; Chemotherapy induced peripheral neuropathy
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcutaneous Acupoints Electrical Stimulation (TAES) group (Experimental): The intervention for TAES group will conduct 2 times per week, total 8 weeks with covering 16 sessions. The intervention will be delivered by a registered nurse with qualified TCM nurse certification. Four bilateral acupoints - Hegu, Shousanli , Zusanli, and Chongyang will be choosen. TAES will be deliveried by electronic acupunture treatment instrument with low frequency. Each session lasts for 60 minutes.
  Interventions: Behavioral: Transcutaneous Acupoints Electrical Stimulation (TAES)
- Sham control group (Sham Comparator): We will adopt a sham control for participants in the sham control group with the same frequency, duration and procedures as the TAES in the experimental group. However, only electrodes will be attached on the four bilateral acupoints, but without any electrical stimulation.
  Interventions: Other: No intervention: sham TAES

INTERVENTIONS:
Behavioral: Transcutaneous Acupoints Electrical Stimulation (TAES) — Transcutaneous Acupoints Electrical Stimulation (TAES) is a kind of physical therapy that use electric current through the electrodes placed on the surface of acupoints to produce clinical effects in the human body.
  Arms: Transcutaneous Acupoints Electrical Stimulation (TAES) group
Other: No intervention: sham TAES — It is designed to look, feel, and be administered identically to the active treatment but lacks its core therapeutic component.
  Arms: Sham control group

SUMMARY:
The first goal of this clinical trial is to assess the feasibility of transcutaneous acupoints electrical stimulation (TAES) on children with acute lymphoblastic leukemia (ALL). The second goal of this clinical trial is to evaluate the preliminary effectiveness of TAES on subject chemotherapy induced peripheral neuropathy (CIPN) symptoms severity, physical function, psychological distress, and quality of life at postintervention and at 1-, and 3-month follow-up postintervention.

The main questions it aims to answer are:

1. What is the feasibility of implementing TAES for children with ALL, as measured by the eligibility rate, consent rate, randomization rate etc.?
2. Does TAES can improve CIPN symptoms severity, physical function, psychological distress, quality of life in children with ALL compared with sham control group?

This proposed research is designed to conduct a two-arm RCT comparing TAES to sham TAES in children with ALL. Subjects in TAES group will receive 8 weeks TAES on four acupoints. Subjects in sham control group will follow the same protocol as the TEAS treatment but with 0 mA, 0 Hz TAES. These two groups will be provided with a leaflet containing self-help materials for CIPN.

ELIGIBILITY:
Inclusion Criteria:

* age between 10 and 17 years old
* diagnosed with ALL
* received neurotoxic chemotherapy
* have developed score 9 or above CIPN symptoms according to Pediatric Chemotherapy-Induced Neuropathy (P-CIN)
* able to communicate and read Chinese

Exclusion Criteria:

* receiving multiple cancer treatment
* had a diagnosis of cancer in the central nervous system cancer, cancer relapse or secondary cancer
* having other neuromuscular disorders, for example, traumatic brain injury and cerebral palsy
* having other systematic diseases that cause toxicity in the peripheral nervous system, such as sickle cell disease (SCD), Guillain-Barre ́ Syndrome (GBS), anterior cutaneous nerve entrapment syndrome (ACNES), obstetric brachial plexus injury (OBPI), type I diabetes mellitus, postherpetic neuralgia (PHN), peroneal nerve injury, and reflex sympathetic dystrophy (RSD)
* acupoints areas with injuries, wounds or allodynia
* participated in any other CIPN non-pharmacological intervention programme
* having any impaired bone marrow suppression
* contraindications to TEAS : such as having a pacemaker, skin infection, damage, or allergy to the electrodes
* suffering from mental illness or using antipsychotic drugs
* parents and children refused to give consent.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility measure - Screening rate | Baseline
  The number of participants being screened divided by the number of participants available for screening
Feasibility measure - Eligibility rate | Baseline
  The number of eligible participants divided by the number of screened participants.
Feasibility measure - Recruitment rate | Baseline
  The number of eligible participants who consent to join divided by the number of eligible participants
Feasibility measure - Randomization rate | Baseline
  The number of consented participants being randomized divided by the number of consented participants
Feasibility measure - Attendance rate | immediately after intervention (T1)
  The number of participants in the experimental group and control group who complete the intervention divided by the number of participants randomized into the group
Feasibility measure - Attrition rate | Baseline, immediately after intervention (T1), 1 month after intervention (T2), and 3 month after intervention (T3)
  The number of participants who drop out divided by the number of participants randomized.
Feasilibility measure - Adverse events | During the study period including 8-week intervention and 3 months follow-up
  It will be denoted as the number of adverse events reported by the participants during the study period.

SECONDARY OUTCOMES:
CIPN severity - Pediatric Chemotherapy-Induced Neuropathy (P-CIN) | Baseline, immediately after intervention (T1), 1 month after intervention (T2), and 3 month after intervention (T3)
  To evaluate the severity of CIPN. The Pediatric Chemotherapy-Induced Neuropathy scale contains 13 items, with eight items to rate CIPN symptoms in the hands and feet and five items to rate the difficulty of performing functional tasks. The total score ranges from 0 to 65 with higher scores indicating more severe CIPN.
Physical functioning - Timed Up and Go test | Baseline, immediately after intervention (T1), 1 month after intervention (T2), and 3 month after intervention (T3)
  Timed Up and Go test (TUG) will be used to evaluate the physical function in children with ALL.
Physical functioning - 30-second sitting-rising test | Baseline, immediately after intervention (T1), 1 month after intervention (T2), and 3 month after intervention (T3)
  30-second sitting-rising test will be used to evaluate the physical function in children with ALL.
Physical functioning - grip strength | Baseline, immediately after intervention (T1), 1 month after intervention (T2), and 3 month after intervention (T3)
  Handheld grip strength meter will be used to evaluate the physical function in children with ALL.
Psychological distress | Baseline, immediately after intervention (T1), 1 month after intervention (T2), and 3 month after intervention (T3)
  National Comprehensive Cancer Network (NCCN) distress thermometer will be used to evaluate the psychological distress of children with leukemia. It included two parts: one is a single-item DT screening tool using an 11-point visual scale for respondents to rate their level of subjective distress from 0 (no distress) to 10 (extreme distress). A cut off value ≥4 was recommended to indicate a distressed patient; another is a 40-items problem list to identify potential sources of distress including practical, family, emotional, physical, and spiritual distress.
Quality of life outcome | Baseline, immediately after intervention (T1), 1 month after intervention (T2), and 3 month after intervention (T3)
  Pediatric Quality of Life Inventory version 3.0 cancer module (PedsQL 3.0 cancer module) will be used to evalute the quality of life for children with leukemia. The scale score was the average of the total item scores, with higher scores representing better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Cancer Hospital of Zhengzhou University, Henan Cancer Hospital, Zhengzhou, China

IPD SHARING:
Plan to Share IPD: No